CLINICAL TRIAL: NCT01535300
Title: Role of Ultrasound Compared to Age-related Formulas for Uncuffed Endotracheal Intubation in a Paediatric Population
Brief Title: Ultrasound and Paediatric Endotracheal Tube Size
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: SonoSite, Inc. (Industry)
Responsible Party: Principal Investigator, Christoph Schramm, M.D., Principal Investigator, Heidelberg University
Other Study IDs: S234/2010
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Uncuffed Endotracheal Intubation
Keywords: Ultrasound; Minimal transverse tracheal diameter; Endotracheal tube size; Paediatric age-based formulas; Sonographic measurement of the trachea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective pediatric surgery
  Interventions: Procedure: Ultrasonography of the trachea

INTERVENTIONS:
Procedure: Ultrasonography of the trachea — Ultrasonographic measurement of the minimal transverse tracheal diameter

SUMMARY:
The aim of the present study was to evaluate the role of ultrasound in paediatric patients to compare the correct size of an uncuffed endotracheal tube (ETT) with the minimal transverse tracheal diameter (MTTD) measured by ultrasound and with tube size predicted by different age-related formulas.

The investigators hypothesize that a prediction of pediatric ETT is possible with the ultrasonographic measurement of the MTTD.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* children <= 5 years of age
* elective surgery requiring endotracheal intubation

Exclusion Criteria:

* missing informed consent
* allergy to ultrasound gel

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children <= 5 years of age scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstanze Plaschke, Professor, Study Chair — Heidelberg University; Christoph Schramm, MD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany